CLINICAL TRIAL: NCT03119896
Title: Supporting Self-management in Chronic Pain: a Collaborative Approach Providing Relevant Tools to Healthcare Professionals and People With Pain.
Brief Title: Supporting Self-management of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Concern (Other)
Collaborators: The Thistle Foundation (Unknown); Health and Social Care Alliance Scotland (the ALLIANCE) (Unknown); Edinburgh and Lothians Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 223092
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Chronic Pain Syndrome; Chronic Pain; Chronic Pain Due to Injury; Chronic Pain Due to Trauma; Chronic Pain Due to Malignancy (Finding); Chronic Pain Post-Procedural; Chronic Pain Hip; Chronic Pain, Widespread
Keywords: chronic pain; self-management; pain management; doctor patient communication; primary care
MeSH Terms: conditions — Chronic Pain; Signs and Symptoms; Agnosia

STUDY DESIGN:
Intervention Model Description: Two groups; one "active group" receiving the intervention, and one "control group" receiving standard care without the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (using Navigator Tool) (Experimental): The participants will receive a copy of the Navigator Tool Intervention, a paper-based information pack including the My Pain Concerns Form, suggested questions to ask your healthcare professional, a goal setting sheet and information on common self-management strategies. They will be encouraged to fill in some of the forms before the consultation, and some during the consultation. They will have consultations with a healthcare professional who has undergone a Self-management Awareness Training with the Thistle Foundation.
  Interventions: Other: The Navigator Tool Intervention
- Control Group (not using Navigator Tool) (No Intervention): These participants will not have access to the Navigator Tool Intervention, and will have consultations with a healthcare professional who has not undergone the Self-management Awareness Training.

INTERVENTIONS:
Other: The Navigator Tool Intervention — The intervention consists of two parts; a training session on self-management of chronic conditions for the healthcare professionals, and a paper-based tool for the patients. Both parts aim to inform and prepare the two parties as to what self-management entails in order to facilitate a constrictive consultation.
  Arms: Intervention Group (using Navigator Tool)

SUMMARY:
Does the Navigator Tool Intervention improve communication regarding self-management during consultations between healthcare professionals and people with chronic pain?

As there is usually no cure for chronic pain, healthcare professionals are increasingly turning to methods of treatment that emphasise management of symptoms rather than elimination of pain. However, as Pain Concern's previous research has shown, there are several barriers to self-management that both healthcare professionals and people with pain face in their consultations in primary care. The Navigator Tool Intervention has been designed to overcome the majority of these barriers through improving the quality of communication regarding self-management during consultations.

In line with the House of Care Model, where care relies on engaged and informed patients, healthcare professionals committed to partnership working, and organisational processes that support this, our intervention prepares both the healthcare professionals and patients for their consultation. By providing a training session for the healthcare professionals in how supported self-management can be brought into the consultation room, and by providing the patients with a paper-based tool that allows them to organise their concerns and questions prior to the consultation, the intervention aims to steer the conversation toward the aspects that the patient needs to discuss in order to better manage their pain.

This study will launch the intervention and evaluate its effectiveness in improving self-management support through conversation. It will be launched over a 3 month period in 4 sites across Scotland; 24 patients will be using the tool with a trained healthcare professional and 24 will act as a control group, receiving standard care without the tool.

Questionnaires assessing the satisfaction with the consultation(s) and communication, as well as confidence in managing one's pain, will be analysed and compared between the two groups. Interviews will be carried out with healthcare professionals and a sample of patients having used the tool to gain a deeper understanding of the usefulness of the intervention and how it may be improved in the future.

DETAILED DESCRIPTION:
This study will involve 4 primary care sites across Scotland, 4-8 healthcare professionals (HCPs) who will administer the intervention, and 48 patient participants (1-2 HCPs and 12 patients at each site). Half of the patient participants will act as the control group and receive no intervention.

4 sites within primary care will be recruited through Pain Concern's current network of healthcare professionals. The sites will consists of general practitioners, physiotherapists and pharmacists, to ensure that the study reflects the usefulness of the intervention across primary care. Each site will nominate 1-2 healthcare professionals who will undergo a training session to learn about supported self-management and how to use the paper-based Navigator Tool effectively. This training will be developed as a collaboration between Pain Concern and the Thistle Foundation, an organisation specializing in supporting self-management for people living with chronic conditions.

Each site will identify 12 patients from their practice who will be asked to participate in the study. With their consent, the patient's contact details will be passed to the researcher who will contact them over the phone and inform them of what the study entails. Prior to this phone call, the patients will have received a written information and a consent sheet through email, post or in person at their practice. The signed consent sheet can be returned the in same way. Once recruited, the participants will be randomly allocated to either the intervention group (24 patients) or the control group (24 patients).

Once allocated to a group, the participant will be sent a pre-intervention pack. There will be two versions of this pack, one for the intervention group and one for the control group. Both packs will contain a Pain Self-Efficacy Questionnaire (PSEQ), and the pack for the intervention group will contain a copy of the Navigator Tool. The participants will be instructed to fill out the questionnaire straight away and return it to the researcher through email or post.

During the active research period (3months), the intervention group will have 2-3 consultations using the tool with a healthcare professional who has undergone the training session. The control group will receive "standard care", i.e. they will not have access to the paper-based tool, and they will be allocated whatever healthcare professional they would have seen if they had not been in the study. There will be no regulation of how many consultations these control participants will have during the research period.

After the 3 month active research period, all patient participants be sent a post-intervention pack. The intervention and control group will be sent identical packs, consisting of a demographics questionnaire, another PSEQ, and a Consultation Quality Index -2 (CQI-2) (which includes the CARE measure).

The scores will be compared between the control and active group and indicate the effect intervention has on our outcome measures. The two most important outcome measures are improvement in communication (measured by CQI-2) and improvement in confidence of pain management (PSEQ). Other outcome measures include engagement with the intervention, perceived participation in decision making, consultations and relational satisfaction and patient-centeredness, extent to which GP was enabling to the patients and perceived efficacy for self-management, scores of which will also be derived from the above questionnaires.

A more in-depth follow-up interview will be conducted with all HCPs and a sample of patient participants (8 patients) spread out over the 4 sites. These interviews will provide a more specific, nuanced and individual understanding of the patients' and healthcare professionals' satisfaction with the intervention and quality of consultations. Possible topics include ease of use, impact on consultation length, effectiveness of communication, required changes to the intervention, and extent to which the intervention achieved aims. These interviews will take place 1-2 months after the last consultation with the tool has taken place, last for around 30-45 minutes, and will be conducted in a venue close to the primary care site the participant was recruited from.

The interviews will be recorded and the researcher will then transcribe the interviews and code them using N-vivo. Themes will be elicited and cross-compared between the participants to establish prevalent experiences, views and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Have experienced pain for more than 3 months

Exclusion Criteria:

* Being unable to communicate in English
* Being unable to attend consultations with a healthcare professional for the duration of the project
* Being currently participating in another research project regarding chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Transcripts of semi-structured interviews with healthcare professionals and patients from Intervention group | Interviews will be carried out 1-2 months after the intervention has finished (the last consultation has taken place).
  Transcripts will be analysed and coded for themes and attitudes, similar concerns and experiences regarding the experience of using the intervention.

SECONDARY OUTCOMES:
Consultation Quality Index - 2 (CQI-2) | Distributed to participants 1 week after the intervention has finished, they will return the filled in questionnaire within 1-2 weeks of having received it.
  Assesses improvement and satisfaction with the communication during consultations. (Patients only)
Pain Self-Efficacy Questionnaire (PSEQ) | First one distributed 1 week before the intervention starts, to be completed and submitted within 1 week. Second will be distributed 1 week after the intervention has ended, to be returned within 1-2 weeks after having received it.
  Assesses improvement to the patients ability to confidently manage their own pain.
CARE measure | Distributed to participants 1 week after the intervention has finished, they will return the filled in questionnaire within 1-2 weeks of having received it.
  Assesses satisfaction with the communication during consultations. (Patients only)

OTHER OUTCOMES:
Transcripts of semi structured interviews with healthcare professionals and patients from the intervention group. | Interviews will be carried out 1-2 months after the intervention has finished (the last consultation has taken place).
  Transcripts will be analysed and coded to elicit attitudes toward strengths and weaknesses of the intervention. It will identify possible improvements and changes to make the intervention easier to use and/or more effective.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela F Bell, MB FFARCSI FFPMCAI FFPMRCA, Principal Investigator — Pain Concern
Locations (5):
- United Kingdom (5):
  - St Margaret's Health Centre, Auchterarder, Scotland
  - Whitesands Medical Practice, Dunbar, Scotland
  - St Triduana's Medical Practice, Edinburgh, Scotland
  - Milngavie Clinic, Milngavie, Scotland
  - Muirhead Medical Centre, Muirhead, Scotland

IPD SHARING:
Plan to Share IPD: No